CLINICAL TRIAL: NCT03718195
Title: Evaluate the Acceptability (Including Gastro Intestinal Tolerance and Compliance) of a Paediatric Tube-feed Formula Ingredients Derived From Real Food for Children Over 12 Months of Age
Brief Title: Acceptability, Gastro Intestinal Tolerance Compliance of a Paediatric Tube-feed Formula Derived From Food for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BLEND001
Record Dates: First submitted 2018-08-22; First posted 2018-10-24 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2018-10

CONDITIONS: Child Nutrition Disorders
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric formula (Other): Each child will receive a new formula for a period of seven days. The new formula is a nutritionally complete standard enteral tube feed, with ingredients derived from real food. The formula is a food for special medical purposes for use under medical supervision.
  The dietitian will determine the feeding regimen on an individual basis and the enteral formula will be provided via a feeding tube
  Interventions: Other: Pediatric Formula

INTERVENTIONS:
Other: Pediatric Formula — One week intake diary, one week tolerance diary, product intake

SUMMARY:
This is an acceptability study to evaluate the gastrointestinal tolerance and compliance over a seven-day period, of pediatric formula for the dietary management of participants with short bowel syndrome; intractable malabsorption; preoperative preparation of undernourished patients; inflammatory bowel disease; total gastrectomy; dysphagia; bowel fistulae; feeding intolerances, developmental disabilities, disease related malnutrition The acceptability data from 15 participants will be collected in order to submit an application to the Advisory Committee on Borderline Substances (ACBS).

DETAILED DESCRIPTION:
Patients well established and stable on a standard enteral tube feed will be changed to a paediatric formula for a period of seven days. This group will act as their own controls. Each child will receive for a period of seven days the paediatric formula, a nutritionally complete standard enteral tube feed.

The dietitian will determine the feeding regimen on an individual basis and the enteral formula will be provided via a feeding tube. A baseline questionnaire will be completed by the dietitian to ensure eligibility of study, current stool patterns or symptoms, current oral intake and weight at the start of the study.

The parents will complete a week intake chart to monitor how much feed has been consumed each day and a tolerance diary to review gastrointestinal symptoms at the start and end of the study.

ELIGIBILITY:
Inclusion Criteria

* Require a tube feed (taking >75% of energy needs from their feeding tube) as part of their dietary management for disease related malnutrition
* Paediatrics aged 1 year above.
* Patients well established and stable on a standard or peptide enteral formula (no gastrointestinal intolerances on current formula)
* Willingly given, written, informed consent from patient or parent/guardian.
* Willingly given, written assent (if appropriate).

Exclusion Criteria

* Inability to comply with the study protocol, in the opinion of the investigator
* Known food allergies to any ingredients (see ingredients list)
* Patients with significant renal or hepatic impairment
* Change in current medication or use of additional macro/micronutrient supplements during the study period, unless clinically indicated and prescribed by the investigator (must be recorded in patient case record file).
* Participation in another interventional study within 2 weeks of this study

Ages: 1 Year to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | Day 7 from baseline
  Incidence of gastrointestinal adverse effects. Tolerance will be evaluated on the basis of the number of gastrointestinal events including diarrhea, constipation, bloating, distension, nausea, vomiting, burping, flatulence and regurgitation and abdominal discomfort or pain reported for subjects during their participation in the study.
Participant compliance | Day 7 from baseline
  Volume of test product prescribed versus actually taken

SECONDARY OUTCOMES:
Body Weight | Day 7 from baseline
  Weight will be measured in Kg

CONTACTS AND LOCATIONS:
Overall Officials: Clare Thornton-Wood, BSc, Principal Investigator — Dietitian
Locations (3):
- United Kingdom (3):
  - Evelina Childrens Hospital, London
  - Chelsea and Westminster Hospital, London
  - East Oxford Health Centre, Oxford

IPD SHARING:
Plan to Share IPD: No